CLINICAL TRIAL: NCT03575585
Title: Maximizing the Patient-counselor Relationship to Reduce Sexual Risk
Brief Title: BEing Safe in Treatment
Acronym: BEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mary Hatch-Maillette, Principal Investigator, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 48767; 5R01HD078163 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Risk Behavior; Sex, Unsafe; Substance Use; Risk Reduction
Keywords: HIV; Counselor Skills Training; Behavioral Intervention; Personalized Feedback Report
MeSH Terms: conditions — Risk-Taking; Unsafe Sex; Substance-Related Disorders; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: This is a 2 x 2 nested factorial design clinical trial. Counselors were randomized to 1) Standard training [2 hours on using a BEST feedback report] or 2) Enhanced training [Standard + 8 hours on discussing sexual risk with patients + monthly coaching]. Patients of participating counselors completed the BEST assessment and were randomized to receive no feedback or a personalized BEST feedback report, and were followed up at 3-, and 6-months (patients). Counselors were assessed at baseline, post-training and 3-months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Comparator: No Feedback, Standard Counselor (Experimental): Patient assigned to a Standard Training counselor, completed the BEST assessment, but did NOT receive a feedback report.
  Interventions: Behavioral: BEST assessment only; Behavioral: Standard Counselor Training
- Active1: Feedback, Standard Counselor (Experimental): Patient assigned to a Standard Training counselor, completed the BEST assessment, and received a personalized feedback report.
  Interventions: Behavioral: BEST assessment plus feedback report; Behavioral: Standard Counselor Training
- Active2: No feedback, Enhanced Counselor (Experimental): Patient assigned to a Enhanced Training counselor, completed the BEST assessment, but did NOT receive a feedback report.
  Interventions: Behavioral: BEST assessment only; Behavioral: Enhanced Counselor Training
- Active3: Feedback, Enhanced Counselor (Experimental): Patient assigned to a Enhanced Training counselor, completed the BEST assessment, and received a personalized feedback report.
  Interventions: Behavioral: BEST assessment plus feedback report; Behavioral: Enhanced Counselor Training

INTERVENTIONS:
Behavioral: BEST assessment only — Patients complete the BEST assessment, a self-report measure containing questions about patients' substance use, sexual risk behaviors, and partner risk levels.
  Other Names: No Feedback
  Arms: Active2: No feedback, Enhanced Counselor; Comparator: No Feedback, Standard Counselor
Behavioral: BEST assessment plus feedback report — Patients complete the BEST assessment, a self-report measure containing questions about patients' substance use, sexual risk behaviors, and partner risk levels. Based on their responses they also receive a personalized feedback report that .provides individualized risk levels in five behavior domains: 1) number of partners, 2) riskiness of partners, 3) condom use, 4) riskiness of sex acts, and 5) sex under the influence of drugs or alcohol.
  Other Names: Feedback
  Arms: Active1: Feedback, Standard Counselor; Active3: Feedback, Enhanced Counselor
Behavioral: Standard Counselor Training — 2 hours of training on how to use the BEST patient feedback report
  Other Names: Standard Training
  Arms: Active1: Feedback, Standard Counselor; Comparator: No Feedback, Standard Counselor
Behavioral: Enhanced Counselor Training — Standard training (2 hrs) plus 8 additional hours (4 modules) of motivation/skills training on a) talking about sex with patients, b) basics of using Motivational Interviewing techniques to review a feedback report, c) teaching patients problem solving skills, and d) teaching patients relationship communication skills.
  Other Names: Enhanced Training
  Arms: Active2: No feedback, Enhanced Counselor; Active3: Feedback, Enhanced Counselor

SUMMARY:
Prior research has shown that many individuals with substance use disorders engage in HIV/sexual risk behaviors, and could strongly benefit from HIV prevention interventions that were delivered as part of their substance abuse treatment. However, discussions about sexual risk are not occurring at an appropriate frequency in treatment settings. This project will test the effects of counselor training and coaching, combined with a brief assessment and feedback tool, on counselor-patient communication about sex and on patient sexual risk behavior.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to substance use disorder treatment in the prior 45 days,
* Age 18 years or older
* Plan to remain in the local area for the next three months
* Assigned to a treatment counselor enrolled in the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Patient unprotected sexual occasions | 3-month follow-up
  Number of unprotected sexual occasions, measured via self-report on the BEST assessment for the prior 90 days
Patient unprotected sexual occasions | 6-month follow-up
  Number of unprotected sexual occasions, measured via self-report on the BEST assessment for the prior 90 days
Discussions of sex during counseling session | 3-month follow-up
  Patient report of number of counseling sessions in past 90 days in which sexual risk was discussed with patients

SECONDARY OUTCOMES:
Patient sexual partners | 3- and 6-month follow-up
  Self-reported number of sexual partners in the 90 days prior to 3- and 6-month follow-up.
Patient unprotected sexual occasions with a casual partner | 3- and 6-month follow-up
  Self-reported number of unprotected sexual occasions with a partner who is not a committed monogamous partner, in the 90 days prior to 3- and 6-month follow-up.
Combining sex and drugs | 3- and 6-month follow-up
  Patient self-report of number of occasions combining drug use and sex in the 90 days prior to 3- and 6-month follow-up.
Patient attitudes toward condoms | 3- and 6-month follow-up
  The Condom Barriers Scale (CBS) (Doyle, Calsyn & Ball, 2009; St. Lawrence et al., 1999) completed by patient participants is a self-report instrument consisting of 29 items worded as short statements and rated by participants on a 5-point Likert-type scale from 1 (strongly agree) to 5 (strongly disagree). Items reflect attitudes about condoms, which may act as barriers towards condom use. Scores are obtained on four conceptual domains: Partner Barriers (8 items), Effects on Sexual Experience (7 items), Access/Availability (8 items), and Motivational Barriers (6 items) and Total Score.
Patient HIV transmission knowledge | 3- and 6-month follow-up
  Patients' HIV knowledge was assessed via self-report using the 18-item HIV Knowledge Questionnaire (HIV-KQ-18: Carey & Schroder, 2002). Items, such as "A woman can get HIV if she has anal sex with a man," are answered "true," "false," or "don't know." Scores range from zero to 18.
Patient risk reduction activities | 3- and 6-month follow-up
  Self-report of engagement in lifestyle risk reduction activities in the 90 days prior to 3- and 6-month follow-up, assessed via the Lifestyle Enhancement Survey. The Lifestyle Enhancement Survey (Calsyn, unpublished), was designed to assess the degree to which patient participants were using strategies to avoid sexual risk and to disentangle their sexual behavior from substance use. Originally designed for a prior pilot study, the version used for this study was modified to align with suggestions included in the Personalized Feedback Report.
Counselor sexual attitudes | Baseline to 1-week post-training and 3-months
  To assess change in counselor sexual attitudes, we used 20 items of the 25-item Sexual Attitude Scale (Hudson, Murphy & Nurius, 1983), an instrument intended to measure the extent to which a participant "adheres to a liberal or a conservative orientation toward human sexual expression" (Hudson et al., 1983, pp. 258). On a 5-point scales, ranging from "Strongly Disagree" to "Strongly Agree," participants rate items, such as "I think there is too much sexual freedom given to adults these days." To reduce participant burden, we abbreviated the scale, removing 5 of 20 items. Two additional items were slightly revised to update language.
Counselor self-efficacy for discussing sex | Baseline to 1-week post-training and 3-month follow-up
  The Sexual Intervention Self-Efficacy Scale (Miller & Byers, 2008) used 16 items via 4 subscales: Comfort/Bias Self-Efficacy (4 items; e.g., I will be able to treat clients with sexual problems even when I don't necessarily agree with their decisions/actions), Skill Self-Efficacy (5 items; e.g., I am unfamiliar with the techniques used to intervene with individuals who have sexual concerns/problems), and Confidence in Ability to Relay Accurate Information (7 items; e.g., I am confident that I can relay accurate information to clients about sexual orientation/identity issues). We also included 3 of 4 items from Miller & Byers (2008; 2012) Willingness to Treat Sexual Issues Scale (e.g., If a couple told me that they were having a sexual problem I would refer them to another clinician). Items were on a 6-point scale ("Strongly Disagree" to "Strongly Agree"). Total scale score equaled the mean of all items. Scoring (after some item reversal) is toward greater self-efficacy.
Counselor skill for discussing sexual issues in counseling sessions | 1-week post-training and 3-month follow-up
  Demonstrated skills in reviewing a personalized feedback report with a Standardized Patient, as coded by independent coders.
Counselor HIV transmission knowledge | Baseline to 1-week post-training and 3-month follow-up
  Counselors' HIV knowledge was assessed via self-report using the 18-item HIV Knowledge Questionnaire (HIV-KQ-18: Carey & Schroder, 2002). Items, such as "A woman can get HIV if she has anal sex with a man," are answered "true," "false," or "don't know." Scores range from zero to 18.

IPD SHARING:
Plan to Share IPD: Yes
The investigative team will make available copies of the BEST survey items, pseudocode for the BEST feedback report, and the counselor training curriculum to other researchers wanting to evaluate their usefulness. Data for this project will consist of quantitative data from patient and counselor assessments. We plan to make the data available to other researchers using two data sharing methods suggested by the NIH Data Sharing Policy brochure. First, we plan to publish information on processes and findings in a timely manner in appropriate peer- reviewed journals that are available online or through requests for copies made directly to the author(s). We will also respond to data requests made directly to the Principal Investigators by removing all identifying information from the data and making them available on a CD-ROM or by posting them on a secure web site. These data will be available at the end of the project after our primary outcome paper is published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available at the end of the project after our primary outcome paper is published.
Access Criteria: Requests can be made to the Principal Investigators.

REFERENCES:
- [Derived] Hatch MA, Wells EA, Masters T, Beadnell B, Harwick R, Wright L, Peavy M, Ricardo-Bulis E, Wiest K, Shriver C, Baer JS. A randomized clinical trial evaluating the impact of counselor training and patient feedback on substance use disorder patients' sexual risk behavior. J Subst Abuse Treat. 2022 Sep;140:108826. doi: 10.1016/j.jsat.2022.108826. Epub 2022 Jun 16. PMID 35751944